CLINICAL TRIAL: NCT06902597
Title: Association Between Sarcopenia And Diabetic Neuropathy In Adults With Type 1 Diabetes, A Pilot Study
Acronym: SARCO_DM1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 7119
Record Dates: First submitted 2025-01-31; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type 1 Diabetes (Experimental): Subjects with type 1 diabetes who will be evaluated for sarcopenia, evaluating body composition through DEXA and muscular strength by handgrip.
  Interventions: Procedure: Dual energy X-ray absorptiometry

INTERVENTIONS:
Procedure: Dual energy X-ray absorptiometry — Very low radiation dose technique to show fat mass (FM) and lean mass (LM)
  Other Names: DEXA (Dual X-ray Absorptiometry)

SUMMARY:
Monocentric interventional prospective study to evaluate the prevalence of sarcopenia in adults with type 1 diabetes (T1DM) and to evaluate the association between diabetic neuropathy and sarcopenia in subjects with T1DM; to evaluate the prevalence of dynapenia in adults with T1DM and its association with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80 years, both sexes
2. Diagnosis of T1DM for at least 10 years, in both multiple daily injections of insulin (MDI) and continuous subcutaneous insulin infusion (CSII)
3. Informed consent before any study activity
4. Ability to fully perform all protocol activities

Exclusion Criteria:

1. Previous diagnosis of T2DM
2. Previous diagnosis of dementia
3. Presence of heart failure (NYHA class III and IV)
4. Presence of muscular disease
5. Diagnosis of neurodegenerative disease (e.g. multiple sclerosis, Parkinson's disease)
6. eGFR evaluated through CKD-EPI formula <20 ml/min /1.73m2 , estimated on previous creatinine dosage
7. Previous history of stroke or cerebrovascular disease
8. Diagnosis of coeliac disease
9. Diagnosis of chronic inflammatory bowel disease
10. Untreated hypothyroidism or hyperthyroidism or not well controlled hypothyroidism or hyperthyroidism with current therapy (TSH >5 or TSH <0.15)
11. Alcohol abuse or consumption of more than 14 alcoholic units weekly
12. Active cancer or therapy
13. Pregnancy
14. Primary hyperparathyroidism
15. Corticosteroid and/or estrogen-progestogen therapy for at least 12 months in medical history
16. On going treatment with antiretroviral therapy
17. On going treatment with immunosuppressive therapy, e.g. cyclosporine, tacrolimus
18. On going treatment with anti-epileptic drugs

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sarcopenia | through study completion, an average of 1 year
  Prevalence of sarcopenia in adult population with T1DM. Sarcopenia will be defined according to the 2018 European Working Group on Sarcopenia in Older People (EWGSOP) guidelines

SECONDARY OUTCOMES:
Prevalence of microvascular complications in subjects with T1DM and sarcopenia | through study completion, an average of 1 year
  Prevalence of peripheral diabetic neuropathy, autonomic diabetic neuropathy, diabetic retinopathy, diabetic nephropathy in subjects with T1DM and sarcopenia
Prevalence of dynapenia | through study completion, an average of 1 year
  Prevalence of dynapenia

CONTACTS AND LOCATIONS:
Overall Officials: Dario Pitocco, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS; UOC Diabetologia, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No